CLINICAL TRIAL: NCT05010811
Title: Two Cases of Pulmonary Cysticercosis Manifesting as Pleural Effusion: Case Report and Literature Review
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-122
Record Dates: First submitted 2021-07-11; First posted 2021-08-18 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2016-09

CONDITIONS: Cysticercosis
Keywords: Cysticercosis; pleural effusion; pulmonary
MeSH Terms: conditions — Cysticercosis; Pleural Effusion

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Isolation lung cysticercosis reports are rare in literature. Most lung lesions were characterized by nodules. The investigators access one case which was characterized with pulmonary cavity and pleural effusion by Gupta N, et al in 2015 from PUBMED and Medline. But pleural effusion and exudative lesions is reported for the first time.

DETAILED DESCRIPTION:
Cysticercosis is an important public health problem in developing countries. The major involvement sites are the central nervous system and the eyes，although striated muscles and subcutaneous tissues are frequently involved in the disseminated form of disease. Pulmonary involvement in cysticercosis is very rare and ill-defined nodular shadows distributed throughout the lung is the usual radiological presentation. Only one case of cysticercosis presenting as lung cavity with pleural effusion has been reported so far in literature. The investigators describe two cases in which pleural effusion due to cysticercosis were detected on X and CT.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of Pulmonary Cysticercosis。
2. With pleural effusion

Exclusion Criteria:

1.No cysticercosis was found by biopsy or antibody test

Ages: 45 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Two patients with pleural effusion presenting with chest tightness and chest pain were enrolled in this study with a definitive diagnosis of cysticercosis confirmed by pleural effusion examination
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2016-10-22 (Actual); Primary Completion 2017-01-18 (Actual); Study Completion 2017-04-28 (Actual)

PRIMARY OUTCOMES:
Amount of pleural effusion | 9 months
  cm
Rate of Eosinophil ratio | 9 months
  Percentage（%）
Changes of lesions under chest radiography or CT | 9 months
  no change, change, complete absorption

CONTACTS AND LOCATIONS:
Overall Officials: Pingli Wang, MD, Study Director — the same research center

IPD SHARING:
Plan to Share IPD: No